CLINICAL TRIAL: NCT04932642
Title: The Effects of Two Different Orders of Concurrent Training on the Interindividual Variability of Health Markers of Metabolic Syndrome and Fitness in Severe/Morbidly Obesity Women. A Randomized Control Trial
Brief Title: Nonresponders by the Session Order Factor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cristian Alvarez (Other)
Collaborators: Universidad de La Frontera (Other)
Responsible Party: Sponsor-Investigator, Cristian Alvarez, Associate Professor, Universidad de Los Lagos
Organization: Universidad de Los Lagos (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RP08042020
Record Dates: First submitted 2021-06-02; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Morbid Obesity; Sports Physical Therapy
Keywords: Morbid obesity; Exercise training; Metabolic syndrome; Concurrent training; Exercise order
MeSH Terms: conditions — Obesity, Morbid; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: We will compare a concurrent training group (HIIT+RT) with morbid obesity with another experimental group of concurrent training with morbid obesity, but with another exercise order (RT+HIIT).
Who Masked: Participant, Investigator
Masking Description: According to availability and the feasibility of the enrolment's requirements, patients will be allocated to aHIIT+RT group with morbid obesity, or to another exercise group of RT+HIIT with morbid obesity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training plus resistance training (HIIT+RT) (Experimental): The HIIT+RT group, the HIIT section consisted of 60 seconds of maximum intensity exercise using a magnetic resistance static bicycle (OxfordTM Fitness, model BE-2701, Chile), followed by 60-120 seconds of passive recovery over the bicycle totally off. This was repeated four to seven times according to the weekly schedule. The intensity of the exercise was measured on the Borg scale of 1 to 10 of perceived exertion and the participants worked at a level of between 6 to 9 points. Second, in the RT section, three to out of four RT exercises were included (according to the planning week), targeting the following different muscle groups: (1) forearm, (2) knee flexors and extensors, (3) trunk, (4) chest, (5) shoulder elevators, (6) horizontal shoulder flexors, (7) extensors, and finally (8) plantar flexors. These exercises were performed in three 3 sets of as many repetitions as possible in 60 seconds, followed by 60 to 120 seconds of passive recovery.
  Interventions: Behavioral: HIIT+RT experimental group
- Resistance training plus High-intensity interval training (RT+HIIT) (Experimental): Firstly, in the RT section, three to out of four RT exercises were included (according to the planning week), targeting the following different muscle groups: (1) forearm, (2) knee flexors and extensors, (3) trunk, (4) chest, (5) shoulder elevators, (6) horizontal shoulder flexors, (7) extensors, and finally (8) plantar flexors. These exercises were performed in three 3 sets of 60 seconds, followed by 60 to 120 seconds of passive recovery, as previously reported. Secondly, in the HIIT+RT group, the HIIT section consisted of 60 seconds of maximum intensity exercise using a magnetic resistance static bicycle (OxfordTM Fitness, model BE-2701, Chile), followed by 60-120 seconds of passive recovery over the bicycle totally off. This was repeated four to seven times according to the weekly schedule. The intensity of the exercise was measured on the Borg scale of 1 to 10 of perceived exertion and the participants worked at a level of between 6 to 9 points.
  Interventions: Behavioral: RT+HIIT experimental group

INTERVENTIONS:
Behavioral: HIIT+RT experimental group — Each experimental group will be compared with their another contrast order session group
  Arms: High-intensity interval training plus resistance training (HIIT+RT)
Behavioral: RT+HIIT experimental group — Each experimental group will be compared with their another contrast order session group
  Arms: Resistance training plus High-intensity interval training (RT+HIIT)

SUMMARY:
Concurrent training (CT, characterised by the inclusion of two exercise modalities), is recognised to improve metabolic syndrome (MetS) markers, but little is known about order session effect on interindividual variability. The purpose of the present study was to describe the effects, and the interindividual variability, of 20 weeks of CT in different order at (i.e., high intensity interval training (HIIT) plus resistance training (RT), compared with another group doing RT plus HIIT) in women with severe/morbidly obesity at risk of MetS.

DETAILED DESCRIPTION:
Morbid obesity, defined as a body mass index (BMI) of 40 kg/m2 (class III obesity), is a chronic disease with life-threatening cardiometabolic consequences such as elevated blood pressure (systolic [SBP] or diastolic BP [DBP]), fasting plasma glucose (FPG), triglycerides (Tg), and low high-density lipoprotein cholesterol (HDL-c), all summarised as metabolic syndrome (MetS). In this sense, exercise training as resistance training (RT), defined as any exercise that causes voluntary skeletal muscle contraction by using external weights such as dumbbells and metal bars, is a known non-pharmacotherapy strategy for improving muscle strength and functional capacity in obese patients undergoing bariatric surgery. Similarly, high-intensity interval training (HIIT), defined as several and brief bouts of high-intensity effort usually by cycling/running, interspersed by recovery periods ), has produced strong evidence for the improvement of cardiometabolic risk factors for type 2 diabetes mellitus, arterial hypertension, central arterial stiffness and, vascular function, and cardiorespiratory fitness. Thus, in individuals with morbid obesity, for example, exercise training has proven to be effective for inducing clinically significant weight loss (5-10%), and for the reduction of cardiovascular risk, following the standard recommendations for these cohorts prior to bariatric surgical. However, some inconsistencies have been described after CT, which are directly concerned with the 'order' (i.e. starting the CT session with MICT followed by RT, or vice versa) of the CT session. However, little is known about the interindividual variability of exercise training (IVET) in relation to different order sessions of CT in morbidly obese populations and health-related outcomes, such as MetS markers. Briefly, IVET means that some subjects achieve benefits after training, and are termed responders (Rs), while others exhibit a worsened or unchanged response, and that is commonly known termed as nonresponders (NRs).

ELIGIBILITY:
Inclusion Criteria:

* being a candidate for bariatric surgery
* aged between 18 and 60 years
* tobe medically authorised
* with a body mass index (BMI) ≥40 kg/m2 or ≥35 kg/m2
* with additional comorbidities (i.e. diabetes, hypertension, insulin resistance) controlled by pharmacotherapy

Exclusion Criteria:

* having physical limitations preventing the performance of exercise (e.g. restricting injuries of the musculoskeletal system)
* having exercise-related dyspnoea or respiratory alterations
* having chronic heart disease with any worsening in the last month
* adhering to less than 80% of the total interventions (these results were excluded from the statistical analyses)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | Baseline to 20-weeks of concurrent training
  Component of metabolic syndrome risk factors
Waist circumference | Baseline to 20-weeks of concurrent training
  Component of metabolic syndrome risk factors
Systolic blood pressure | Component of metabolic syndrome risk factors
  Component of metabolic syndrome risk factors
Diastolic blood pressure | Baseline to 20-weeks of concurrent training
  Component of metabolic syndrome risk factors
High-density lipoprotein cholesterol | Baseline to 20-weeks of concurrent training
  Component of metabolic syndrome risk factors
Triglycerides | Baseline to 20-weeks of concurrent training
  Component of metabolic syndrome risk factors

SECONDARY OUTCOMES:
Body mass (kg) | Baseline to 20-weeks of concurrent training
  Anthropometry parameter related with health and intervention effects. This outcome will be measured by a bio-impedance scale (TANITATM, model 331, Tokyo, Japan).
Body mass index (height/m2) | Baseline to 20-weeks of concurrent training
  Anthropometry parameter related with health and intervention effects
Body fat percentage (%) | Baseline to 20-weeks of concurrent training
  Anthropometry parameter related with health and intervention effects
Body fat (kilograms) | Baseline to 20-weeks of concurrent training
  Anthropometry parameter related with health and intervention effects
Skeletal muscle mass (kg) | Baseline to 20-weeks of concurrent training
  Body composition parameter related with health and intervention effects. This outcome will be measured by a bio-impedance scale (TANITATM, model 331, Tokyo, Japan).
Lean mass (kg) | Baseline to 20-weeks of concurrent training
  Body composition parameter related with health and intervention effects. This outcome will be measured by a bio-impedance scale (TANITATM, model 331, Tokyo, Japan).
Total cholesterol | Baseline to 20-weeks of concurrent training
  Metabolic parameter related with health and intervention effects
Low-density lipoprotein cholesterol | Baseline to 20-weeks of concurrent training
  Metabolic parameter related with health and intervention effects
Handgrip muscle strength (kg) | Baseline to 20-weeks of concurrent training
  Physical fitness outcome related with health and intervention effects. This outcome will be measure using a digital dynamometer (BaselineTM Hydraulic Hand Dynamometers, USA),
Six minutes walking test | Baseline to 20-weeks of concurrent training
  Physical fitness outcome related with health and intervention effects

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Alvarez, PhD, Study Director — Universidad de Los Lagos
Locations (1):
- Cristian ALvarez, Osorno, Llanquihue, Chile

IPD SHARING:
Plan to Share IPD: No
The participant's information will be available by e-mail according to with researcher's requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04932642/Prot_SAP_000.pdf